CLINICAL TRIAL: NCT03874910
Title: Pathology Analysis of OPMD Patient Myotomies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0115-18-HYMC
Record Dates: First submitted 2019-03-04; First posted 2019-03-14 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Oculopharyngeal Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Oculopharyngeal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to characterize the effect of OPMD mutation on muscle function. Muscle samples will be received from oculopharyngeal muscular dystrophy (OPMD) patients who undergo cricopharyngeal muscle-cutting surgery, as part of their routine healthcare and treatment.

ELIGIBILITY:
Inclusion Criteria:

* OPMD patients both male and female.
* OPMD patients between the ages 18-70 years.
* OPMD patients who are referred to the cricopharyngeal muscle-cutting surgery as part of their usual treatment.

Exclusion Criteria:

• OPMD patients not referred to the cricopharyngeal muscle-cutting surgery as part of their usual treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who suffer from oculopharyngeal muscular dystrophy (OPMD).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-03-19 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Number of genes that show changes in RNA profile, measured by sequencing. | Data will be collected within four years.
  RNA profile analysis of OPMD muscle samples will be compared to unaffected muscle samples using sequencing to identify gene numbers.
Number of genes that show changes in protein profile, measured by SDS page. | Data will be collected within four years.
  Protein profile analysis of OPMD muscle samples will be compared to unaffected muscle samples to identify gene numbers using SDS page.

CONTACTS AND LOCATIONS:
Overall Officials: Itzhak Braverman, Doctor (MD), Principal Investigator — Hillel Yaffe Medical Center, Israel
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel